CLINICAL TRIAL: NCT00891709
Title: A Phase 1, First in Man, Safety, Tolerability and Pharmacokinetic Study of Single Ascending and Multiple Cutaneous Doses of LEO 29102 2.5 mg/g Cream or LEO 29102 Cream Vehicle in Healthy Male Subjects
Brief Title: LEO 29102 Single and Multiple Dose Study by Dermal Application
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LEO 29102-C01
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2010-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — 2-(6-(2-(3,5-dichloro-4-pyridyl)acetyl)-2,3-dimethoxyphenoxy)-N-propylacetamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): LEO 29102 2.5 mg/g cream
  Interventions: Drug: LEO 29102
- 2 (Placebo Comparator): LEO 29102 cream vehicle
  Interventions: Drug: LEO 29102

INTERVENTIONS:
Drug: LEO 29102 — First-in-man. Healthy volunteers

SUMMARY:
The principal aim of this study is to obtain safety, tolerability and pharmacokinetic data when LEO 29102 is administered cutaneously as single and multiple doses to healthy male subjects.

The study is divided into one single dose part followed by a multiple dose part.

ELIGIBILITY:
Inclusion Criteria:

* Male adults between the age of 18 and 55 years (both inclusive) and with a BMI between 19 and 30 kg/m2 (both inclusive).
* Subjects must be healthy as determined by medical history, physical examination, electrocardiogram (ECG), blood pressuer and heart rate, and clinical laboratory evaluation.

Exclusion Criteria:

* Subjects who show signs of eczema or other skin lesions.
* Subjects who have any clinical signs of allergic diseases (excluding non active hay fever).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability

SECONDARY OUTCOMES:
To determine the pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Priestley, MBChB MFPM, Principal Investigator — LCG Bioscience, Bourn Hall, Bourn, Cambridgeshire, CB23 2TN, UK
Locations (1):
- LCG Bioscience, Bourn, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No